CLINICAL TRIAL: NCT04506424
Title: High Resolution CT Guided Cochlear Implant Programming
Brief Title: CT Guided CI Programming
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-17575
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Cochlear Implants; Hearing Loss; Amusia
Keywords: Music perception; Place-pitch mismatch; Place coding; Cochlear duct length; Flat panel computed tomography; Cochlear implant programming; Frequency allocation table
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Participants will undergo a Flat Panel (high resolution) CT scan of the temporal bones, including the inner ear structures. The research team will make measurements of the cochleas from the CT scans, including cochlear duct length and depth of CI electrodes. The research team will generate custom frequency allocation tables to be used in the experimental programs for the CI.
  Participants may have the experimental programs uploaded to their CI and use these programs to listen to speech and music stimuli and provide feedback. The participants may be asked to listen to these programs for acute and/or chronic periods of time. Participants may also have their performance on speech and music assessments measured using a clinical default program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT-Based Program for First Year of CI Use (Experimental): The Flat Panel CT scan will take place after a CI has been implanted and prior to the CI device activation.
  The CI device will be activated using a CT-based program. The participant may continue to use this program for 1 year. Speech and music perception abilities will be monitored at regular intervals (approx. at 1, 3, 6, and 12 months post-activation).
  After the 1 year of experimental program use, the participant may be switched over to a program that uses only the clinical default settings for 1 month; after which the participant will again complete the speech and music test battery.
  At the end of the 13 month study the participant may choose whether to use the CT-based program or the clinical default program moving forward.
  Interventions: Other: CT Guided Cochlear Implant Programming

INTERVENTIONS:
Other: CT Guided Cochlear Implant Programming — Flat Panel (high resolution) CT scans of the temporal bones, including the inner ears, will be obtained. The research team will use the scans to generate custom cochlear implant (CI) programs for use by the participants.

SUMMARY:
The current standard of care for cochlear implants (CI) does not address the significant pitch-place mismatch that is inherent in cochlear implantation (see detailed description below). The present study uses postoperative Flat Panel (higher resolution than standard) CT imaging to measure where CI electrodes sit within an individual's cochlea; doing so allows for more accurate frequency mapping (and thus pitch perception). The hypothesis of this study is that long-term (1 year) use of CT image-based frequency maps, beginning on the first day of CI activation, will improve user performance in the areas of speech and music perception, as compared to the use of default programming settings.

DETAILED DESCRIPTION:
Pitch perception is a fundamental component of how humans process sound. Individuals who use cochlear implants (CIs), surgically implanted devices which are able to restore a limited range of hearing, struggle with pitch perception for a variety of reasons. Although CIs can often restore the ability to hear speech from a single talker in quiet, perception of more complex auditory stimuli like music is severely limited. CI users often report music as being difficult, even displeasing, to listen to. These experiences can be immensely frustrating, especially for people who experience deafness later in life and have built strong emotional attachments to music, such as musicians or audiophiles.

Cochlear implant programming (also called "mapping") is done using a set of generally-accepted default settings without taking into account individual differences of precisely where CI electrodes are physically located in the cochlea. For this reason, CI users commonly experience a place-pitch mismatch between the stimulation by an electrode in response to a given frequency and the actual frequency specified by the original cochlear location. CI users vary widely in their ability to adapt to place-pitch mismatch; some adapt completely, others partially, and others not at all. The length of time in which an individual takes to adapt is also highly variable. Bilateral CI users may have differing adaptation between ears, leading to distortion of sound localization and speech in noise perception abilities.

Flat Panel Computed Tomography (FPCT) is an imaging technique that consistently produces high quality images with identification of the delicate cochlear structures and the cochlear implant (CI) electrode contacts. FPCT imaging of the cochlea, combined with 3D curved multiplanar reconstruction (MPR) software, has been shown to yield reliable cochlear duct length measurements. With these resources, measurements of cochlear length and determination of intracochlear electrode location relative to standardized cochlear landmarks can be produced. These data are then utilized to create individualized frequency allocation tables relevant to the actual physical location of CI electrode contacts.

In this study, FPCT imaging, 3D curved MPR, and applied mathematics are used to quantify the difference between theoretical and actual electrode contact placement with respect to pitch-place mapping. Previous results have revealed significant deviations between predicted and programmed characteristic frequencies, which are relevant for accurate speech, pitch, and music perception. The goal of the study is to gather FPCT scans on a cohort of 20 new CI recipients, and characterize the impact of long-term (1 year) personalized pitch-place maps on a battery of speech and music metrics. The performance with the FPCT-based programs will then be compared to performance using the manufacturer default settings.

The novel aspect of this study involves working with newly implanted CI recipients and programming these patients with custom CT-based programs. More specifically, CT-based programs will be given to new CI recipients before any acclimation or programming of clinical default maps occur. This differentiates the study from prior ones, as CT-based programming has only been investigated in populations who have already used clinical default maps for some substantial period of time (e.g. for 3 months, 5 years, etc.). Participants will participate in a series of testing sessions to evaluate their speech and music perception abilities over the course of the study. At the end of the study, participants will be allowed to keep their preferred listening programs (i.e., experimental and/or default program).

The researcher team hypothesizes that bypassing the use of a clinical-based map is imperative to fully understanding the effects of CT-based programming, as those who have already used clinical default programs demonstrate much higher degrees of place-pitch mismatch at baseline. By providing a new CI recipient with a custom CT-based program on their very first day of electrical hearing (CI activation), there is a unique and novel opportunity to minimize pitch-place mismatch from the outset, and to bypass the period of time that the vast majority of CI recipients have when first adapting to a clinical default program.

ELIGIBILITY:
Inclusion Criteria:

* Has or plans to have a MED-EL cochlear implant (CI)
* Has not yet had their CI activated
* Be able and willing to participate in all of the research appointments for follow-up testing (e.g., 1, 3, 6, 12, and 13 months post-CI activation)
* Be willing to use the CI full-time (during waking hours) for 13 months post-activation
* Is able to speak and read American English
* Uses oral/aural communication as primary communication modality

Exclusion Criteria:

* Intra-cochlear electrodes known to be open or short-circuits
* Partially-inserted CI with fewer than 10 intra-cochlear electrodes
* Any concomitant condition(s) that may affect performance on speech and music test battery (e.g., cognitive impairment)
* Atypical cochlear anatomy (e.g., fewer than 2 turns of the cochlea)
* Pregnancy (a contraindication for CT scan)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Change in score on the Consonant-Nucleus-Consonant (CNC) Test between chronic use of the CT-based program (~12 months post-activation) and chronic use of the clinical default program (~1 month post-switchover) | Baseline (12 months post-activation) to 1 month post-switchover (13 months post-activation)
  * The CNC word test consists of lists of monosyllabic (single syllable) words with equal phonemic distribution across lists. There are 50 words per list. Performance is calculated based on percentage of words correct (from 0 to 100) and/or percentage of phonemes correct (from 0 to 100).
  * From CI activation until ~12 months post-activation the participant will use the CT-based program. At that time the participant will "switchover" to the clinical default program, which will be used for ~1 month.

CONTACTS AND LOCATIONS:
Overall Officials: Charles J Limb, MD, Principal Investigator — University of California, San Francisco; Melanie L Gilbert, AuD, Study Director — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data/results from participants of this study will be de-identified prior to publication. Data and materials from this study will be uploaded to the repository provided by the Library of the University of California, San Francisco (Dryad).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data and materials will become available after the corresponding manuscript has completed a peer review process and is accepted for publication.
Access Criteria: Publicly available

REFERENCES:
- [Background] Jiam NT, Pearl MS, Carver C, Limb CJ. Flat-Panel CT Imaging for Individualized Pitch Mapping in Cochlear Implant Users. Otol Neurotol. 2016 Jul;37(6):672-9. doi: 10.1097/MAO.0000000000001060. PMID 27273394
- [Background] Jiam NT, Gilbert M, Cooke D, Jiradejvong P, Barrett K, Caldwell M, Limb CJ. Association Between Flat-Panel Computed Tomographic Imaging-Guided Place-Pitch Mapping and Speech and Pitch Perception in Cochlear Implant Users. JAMA Otolaryngol Head Neck Surg. 2019 Feb 1;145(2):109-116. doi: 10.1001/jamaoto.2018.3096. PMID 30477013